CLINICAL TRIAL: NCT03031145
Title: Investigation of the Impact of Smoking Status on Allergen-induced Nasal Airway Inflammation Using a Cat Hair (Felis Domesticus) Extract Nasal Allergen Challenge Model
Acronym: Kitty Nose
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1686
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Tobacco Smoking; Healthy Participants; E-cigarette Smokers
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Felis Domesticus treated Non-smoker (Active Comparator)
  Interventions: Biological: Felis Domesticus
- Felis Domesticus treated E-cigarette smoker (Active Comparator)
  Interventions: Biological: Felis Domesticus
- Felis Domesticus treated Cigarette smoker (Active Comparator)
  Interventions: Biological: Felis Domesticus

INTERVENTIONS:
Biological: Felis Domesticus — Nasal Administration of Felis Domesticus
  Other Names: Cat Allergen

SUMMARY:
The purpose of this pilot study is to evaluate allergen-induced nasal airway inflammation following nasal application of felis domesticus, or cat, extract in e-cigarette users, cigarette smokers, and non-smokers.

DETAILED DESCRIPTION:
The recent increase in popularity of e-cigarettes for smoking cessation or in combination with conventional cigarettes has let to safety concerns regarding their potential role in respiratory disease. These tobacco alternatives devices were initially perceived as a "safer" alternative to cigarettes and were marketed without much known about their health effects. Increasing evidence that while they contain fewer toxins and carcinogens than conventional cigarettes, they do involve delivery of ultrafine particles to the lower airways and can contain heavy metals and other chemicals. Tobacco Smoke may augment allergic inflammation resulting from allergic rhinitis and/or asthma. Animal models of allergic asthma demonstrate aggravation of allergen -induced airway inflammation following inhalation of e-cig cartridge solution, with increased airway eosinophil infiltration, production of Th2 cytokines, and airway hyperresponsivness. In vitro studies in human tissues have demonstrated pro-inflammatory responses in a similar way as tobacco smoke, yet a head-to-head comparison of the effects of these two exposures has not been performed in humans.

Use of tobacco products remains a pervasive problem in our society and around the world, with significant impact on respiratory health and quality of life. With the emergence of new non-tobacco based nicotine products like e-cigarettes, it is important to understand the impact these substances have on respiratory health and disease. The aim o f this study is to study the impact of these products on allergic inflammation in cat allergic subjects who already routinely use e-cigarettes and to compare their response to those of cigarette smokers and non-smokers. A thorough understanding of the potential health impacts of tobacco alternative substances in seeded, especially given the rising popularity of such products with adolescents and young adults to whom these substances have particular appeals given the purported safety: and variety of flavors to chose from.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-50 years
2. Specific allergy to cat hair Felis domesticus confirmed by positive immediate skin test response
3. Subjects may be enrolled with mild asthma if a Forced Expiratory Volume in 1 second (FEV1) of at least 80% of predicted and a Forced Expiratory Volume in 1 second to Forced Vital Capacity (FVC) ratio (FEV1/FVC ratio) of at least .75 (without use of bronchodilator medications for 12 hours), consistent with lung function of persons with mild episodic or mild persistent asthma is demonstrated. For the purpose of this protocol, an asthmatic individual will be defined as having a) positive methacholine challenge with a provocative concentration of methacholine producing a 20% fall in FEV1 (PC20 methacholine) with less than or equal to 10 mg/ml; OR b) physician diagnosed asthma with symptoms and chronic daily therapy consistent with the mild asthma
4. Ability to withhold antihistamine medications for one week prior to baseline and allergen challenge visits.
5. Subjects must be able and willing to give informed consent.
6. Subjects will be classified as tobacco smokers, e-cigarette users, or non-smokers

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the allergen challenge study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, bleeding disorder, or chronic thyroid disease.
2. Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
3. Use of systemic steroid therapy within the preceding 12 months for treatment of an asthma exacerbation.
4. Use of inhaled or nasal steroids, cromolyn or leukotriene receptor antagonists (Montelukast or Zafirkulast) within the past month (except for use of cromolyn exclusively prior to exercise).
5. Use of allergen immunotherapy.
6. Use of daily theophylline within the past month.
7. Use of nasal medications that might alter the response to nasal allergen challenge including anti-inflammatory and anti-histamine agents within one week of challenge.
8. Inability to withhold inhaled or oral bronchodilator medications for 12 hours prior to allergen challenge.
9. Pregnancy or nursing a baby.
10. Women of child-bearing age who are not using dependable contraception (such as birth control pills, IUD, estrogen patches) or who are not completely abstinent.
11. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
12. Exacerbation of asthma more than 2x/week which would be characteristic of a person with moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
13. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
14. Viral upper respiratory tract infection within 4 weeks of challenge.
15. Any acute infection requiring antibiotics within 4 weeks of challenge.
16. Participating in an allergen inhalation study within 2 weeks of this challenge or use of any investigational agent within the last 30 days.
17. Use of tricyclic antidepressants or beta-blockers.
18. Use of MAO inhibitors or any medications known to interfere with the treatment of anaphylaxis.
19. Subjects with a history of immunologic disease or undergoing immune suppression for cancer or other diseases.
20. Subjects with acute inflammatory conditions in the nose or paranasal sinuses, such as sinusitis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Change in eosinophils/mL in nasal lavage fluid (NLF) | Pre- and 4 hours post- nasal allergen challenge
  NLF will be collected immediately prior to administration of the nasal allergen challenge. 4 hours after administration of a bolus provocative dose of allergen (determined at screening day visit nasal allergen challenge), NLF will be collected. Pre- and 4 hours post-challenge NLF will be analyzed for cellularity. Values will be compared across e-cigarette smokers, tobacco cigarette smokers, and non-smokers.

SECONDARY OUTCOMES:
Nasal lavage fluid cytokines | Pre- and 4 hours post- nasal allergen challenge
  NLF will be collected immediately prior to administration of the nasal allergen challenge, and 4 hours post-nasal allergen challenge. Cytokine levels will be quantified with commercially available ELISAs.
Nasal epithelial cell messenger ribonucleic acid (mRNA) | Baseline (within two months of nasal allergen challenge) and 4 hours post- nasal allergen challenge
  Nasal epithelial cell biopsies will be collected at baseline (within two months of nasal allergen challenge), and 4 hours post-nasal allergen challenge. Gene expression changes will be quantified using qRT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No